CLINICAL TRIAL: NCT06497049
Title: An Open Randomized Study of Comparative Pharmacokinetics and Biosimilarity of GP40221, Solution for Subcutaneous Administration 1.34 mg/ml (GEROPHARM) and Ozempic®, Solution for Subcutaneous Administration 1.34 mg/ml in Healthy Volunteers
Brief Title: Open Randomized Study of Comparative Pharmacokinetics and Biosimilarity of GP40221 (GEROPHARM LLC, Russia) and Ozempic®.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Geropharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GP40221-P4-01-01
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-05

CONDITIONS: Pharmacokinetics; Safety Issues; Bioequivalence
Keywords: semaglutide; ozempic
MeSH Terms: interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: An open randomized study of comparative pharmacokinetics and biosimilarity of GP40221, solution for subcutaneous administration, 1.34 mg/ml and Ozempic®, solution for subcutaneous administration, 1.34 mg/ml in parallel groups in healthy volunteers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GP40221 (Experimental): GP40221 is administered subcutaneously into the subcutaneous fat of the anterior abdominal wall at a dose of 0.5 mg using a pen injector.
  Interventions: Drug: GP40221
- ozempic (Active Comparator): Ozempic® is administered subcutaneously into the subcutaneous fat of the anterior abdominal wall at a dose of 0.5 mg using a pen injector
  Interventions: Drug: ozempic

INTERVENTIONS:
Drug: GP40221 — Solution for Subcutaneous Administration 1.34 mg/ml
  Other Names: semaglutide
  Arms: GP40221
Drug: ozempic — Solution for Subcutaneous Administration 1.34 mg/ml
  Other Names: semaglutide
  Arms: ozempic

SUMMARY:
Study of comparative pharmacokinetics and biosimilarity of drugs containing semaglutide - GP40221 and Ozempic® in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent to participate in the study.
* Males with a verified diagnosis "healthy" according to the data of standard clinical, laboratory and instrumental examination methods.
* Age 18-45 years old inclusive.
* Body mass index 18.5 - 29.9 kg/m2.
* Agree to use an adequate method of contraception (double barrier method) during the entire period of participation in the study and for 3 weeks after its completion.
* Consent to all restrictions imposed during the study.
* Citizenship of the Russian Federation.

Exclusion Criteria:

* Burdened allergic history, drug intolerance.
* Hypersensitivity to heparin, semaglutide and any of the excipients of the study drug.
* Any acute and chronic diseases, incl. but not limited to:

  1. diseases of the cardiovascular, bronchopulmonary, neuroendocrine systems, as well as diseases of the gastrointestinal tract (including diseases of the colon), liver, kidneys, blood;
  2. positive test results for hepatitis C (antibodies) or hepatitis B (surface antigen), HIV (antibodies to HIV-1/2), syphilis (antibodies to Treponema pallidum).
* Deviations from normal values of heart rate (60-80), SBP (100-130 mm Hg), DBP (60-85 mm Hg), NPV (16-20), body temperature (35.7 - 37.0 °C).
* ECG Deviations, according to a specialist, during screening.
* laboratory tests results deviations from the normal values.
* Hard-to-reach veins of the upper extremities, vein thrombosis, thrombophlebitis in a family history of close relatives, "compromised" veins due to frequent previous venipunctures.
* Surgical interventions on the gastrointestinal tract (with the exception of appendectomy) in history.
* Acute infectious diseases less than 4 weeks prior to screening.
* History of medullary thyroid cancer and/or multiple endocrine neoplasia type 2, including family history.
* History of chronic or acute pancreatitis.
* Regular use of any prescription and over-the-counter medications (in particular drugs that reduce heart rate), dietary supplements, vitamins less than 2 weeks before the start of screening, taking St. John's wort (Hypericum perforatum) less than 30 days before the start screening.
* Use of semaglutide or other analogues of human glucagon-like peptide-1 (GLP-1) within 6 months before screening.
* Use of depot injections or implants of any medications 3 months before the start of screening.
* Significant blood loss (more than 450 ml of blood or plasma) within 3 months prior to screening, due to, including, but not limited to, blood donation, blood loss during advanced surgery or trauma.
* Drinking alcohol in quantities exceeding 10 units per week (on average) (1 unit of alcohol is equivalent to 500 ml of beer, 200 ml of dry wine or 50 ml of strong alcoholic drinks) or anamnestic information about alcoholism, drug addiction, abuse of strong drugs.
* Positive test results for alcohol, drug use and the use of strong drugs.
* Nicotine addiction (regular tobacco use, including smoking of all types of electronic cigarettes, hookahs, snuff, etc. less than 6 months prior to screening).
* Participation in a clinical trial of any drugs (including experimental drugs) or experimental medical devices for 3 months or 5 half-lives prior to Screening, whichever is longer.
* Any diet (eg vegetarian, fasting, etc.) or lifestyle (including night work and extreme physical activity such as heavy lifting) that may interfere with the study.
* Taking drugs that have a pronounced effect on hemodynamics, liver function, etc. (barbiturates, omeprazole, cimetidine, etc.) less than 30 days before screening.
* Consumption of citrus fruits (including grapefruit and grapefruit juice), cranberries (juice, fruit drink, etc.), starfruit or pomelo 14 days before the start of screening.
* Incomplete recovery from surgery or surgery scheduled while the volunteer was participating in the study.
* Other diseases/conditions that, in the opinion of the researcher, may affect the pharmacokinetics of the active substance of the drugs or increase the risk to the health of the volunteer.
* Tattoos or piercings less than 30 days before screening.
* Volunteers who are obviously or likely, in the opinion of the investigator, unable to understand and evaluate the information on this study as part of the informed consent process, in particular regarding expected risks and possible discomfort.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — naturaly male
Enrollment: 120 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
AUC 0-t | -60, -30, 0 minutes and 2, 4, 8, 10, 12, 16, 24, 36, 48, 60, 72, 96, 144, 192, 240, 288 hours after injection
  Total area under the "concentration of an active substance - time" curve in the time interval from 0 (the moment of drug administration) to the collection of the last blood sample with a determined concentration of the active substance at time point t
Cmax | -60, -30, 0 minutes and 2, 4, 8, 10, 12, 16, 24, 36, 48, 60, 72, 96, 144, 192, 240, 288 hours after injection
  Maximum concentration of the active substance in the blood plasma of volunteers during the observation period

SECONDARY OUTCOMES:
tmax | -60, -30, 0 minutes and 2, 4, 8, 10, 12, 16, 24, 36, 48, 60, 72, 96, 144, 192, 240, 288 hours after injection
  Time to reach the maximum concentration (Cmax) of an active substance in the blood plasma of volunteers
t1/2 | -60, -30, 0 minutes) and 2, 4, 8, 10, 12, 16, 24, 36, 48, 60, 72, 96, 144, 192, 240, 288 hours after injection
  half-life of an active substance
λz | -60, -30, 0 minutes) and 2, 4, 8, 10, 12, 16, 24, 36, 48, 60, 72, 96, 144, 192, 240, 288 hours after injection
  constant of elimination of an active substance
AUC0-∞ | -60, -30, 0 minutes) and 2, 4, 8, 10, 12, 16, 24, 36, 48, 60, 72, 96, 144, 192, 240, 288 hours after injection
  total area under the "concentration of an active substance - time" curve in the time interval from 0 (the moment of drug administration) to infinity

CONTACTS AND LOCATIONS:
Overall Officials: Sergei Noskov, MD, Pr., Principal Investigator — Yaroslavl State Institution of Healthcare "Clinical Hospital No. 3"
Locations (1):
- Yarosslavl Clinical Hospital #3, Yaroslavl, Russia